CLINICAL TRIAL: NCT03659968
Title: Phase I Dose-escalation Study of Adapted Physical Activity in Children and Adolescent Suffering From Advanced Malignancies.
Brief Title: Initiation of Adapted Physical Activity for Patients With Advanced Pediatric Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-70
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXPERIMENTAL GROUP (Experimental): patients in advanced phase of pediatric cancer Physical activity training will be performed in drug development
  Interventions: Other: Physical activity training

INTERVENTIONS:
Other: Physical activity training — brisk walking on treadmill and exercises of muscular strengthening with varying durations and intensities depending on physical capabilities of patients

SUMMARY:
Adapted physical activity (APA) in the context of cancer is a field of growing interest and has been explored in numerous publications. In adults, the effects of APA on survival, symptoms and quality of life are established and its physiological consequences on immunity, angiogenesis and hormone secretion are under investigation.

In children and adolescents, evidence is scarce: pilot studies show clinical benefit of physical activity practiced in a wide variety of situations and protocols with low level of scientific evidence. It is therefore not possible to recommend this practice in pediatrics despite the large number of initiatives and the conviction of many clinicians that there is a benefit for patients. In particular, there are few trials in children with advanced cancer pathologies or in palliative care. However, these patients have a high prevalence of severe symptoms (pain, digestive disorders, asthenia, and anxiety) for which physical activity may represent a therapeutic option.

The purpose of our study is to describe a protocol of adapted physical activity and to evaluate its feasibility and toxicity according to a well-known and validated methodology in oncology used in drug development.

Methodology is based on a simple and reproducible intervention combining brisk walking on treadmill and exercises of muscular strengthening with varying durations and intensities depending on physical capabilities of patients.

The primary objective is to define the volume of physical activity that can be proposed to a patient starting APA based on the assessment of his physical condition evaluated by a 6-minutes walking distance test.

Inclusion criteria are broad to allow study population to represent the diversity of patients in pediatric palliative oncology. Stratification of patients in three groups based on a 6-minutes walking distance test aims to adapt intervention to physical capability of patients and improve tolerance.

Dose escalation will be set with a "3 + 3" regimen used in drug early phases trials.

Primary outcome measure is perceived tolerance evaluated by the patient with a subjective scoring on CREST scale. Any score greater than 8/10 defines intolerance.

DETAILED DESCRIPTION:
Adapted physical activity (APA) in the context of cancer is a field of growing interest and has been explored in numerous publications. In adults, the effects of APA on survival, symptoms and quality of life are established and its physiological consequences on immunity, angiogenesis and hormone secretion are under investigation.

In children and adolescents, evidence is scarce: pilot studies show clinical benefit of physical activity practiced in a wide variety of situations and protocols with low level of scientific evidence. It is therefore not possible to recommend this practice in pediatrics despite the large number of initiatives and the conviction of many clinicians that there is a benefit for patients. In particular, there are few trials in children with advanced cancer pathologies or in palliative care. However, these patients have a high prevalence of severe symptoms (pain, digestive disorders, asthenia, and anxiety) for which physical activity may represent a therapeutic option.

The purpose of our study is to describe a protocol of adapted physical activity and to evaluate its feasibility and toxicity according to a well-known and validated methodology in oncology used in drug development.

Methodology is based on a simple and reproducible intervention combining brisk walking on treadmill and exercises of muscular strengthening with varying durations and intensities depending on physical capabilities of patients.

The primary objective is to define the volume of physical activity that can be proposed to a patient starting APA based on the assessment of his physical condition evaluated by a 6-minutes walking distance test.

Inclusion criteria are broad to allow study population to represent the diversity of patients in pediatric palliative oncology. Stratification of patients in three groups based on a 6-minutes walking distance test aims to adapt intervention to physical capability of patients and improve tolerance.

Dose escalation will be set with a "3 + 3" regimen used in drug early phases trials.

Primary outcome measure is perceived tolerance evaluated by the patient with a subjective scoring on CREST scale. Any score greater than 8/10 defines intolerance.

Secondary objectives include the description of tolerance during sessions with shortness of breath and pain scores, the comparison of objective (HR) and perceived measures, and the study of patient's characteristics and medical history as confusion factors.

The evolution of the patient's physical capability will be evaluated at the end of the study. The continuation of physical activity beyond the duration of participation will be documented. The impact on pathology-related symptoms and quality of life will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 5 to 17 years old.
* Cancer with no curative therapeutic options.
* Stable disease (with or without treatment).
* Ability to complete 100 meters walking without help and muscular strengthening exercises.
* Written informed consent, including agreement of parents or legal guardian for minors.

Exclusion Criteria:

* Participation to another Phase I trial
* Dyspnoea exertional
* Cardio-vascular pathology
* Life expectancy of less than 3 months
* Progressive disease
* Expected inability to comply to medical follow up

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Perceived tolerance | 6 weeks
  Evaluated by the patient with a subjective scoring on scale (from 0 to 10). Any score greater than 8/10 define intolerance. Any score under 8/10 definite "acceptable tolerance"

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assiatnce Publique Des Hopitaux de Marseille, Marseille, PACA, France